CLINICAL TRIAL: NCT03233607
Title: Optimal Time for Postpartum Hemoglobin Assessment and Its Correlation With Estimated Blood Loss (EBL)/Quantitative Blood Loss (QBL)
Brief Title: Time of Postpartum Hemoglobin Assessment and Blood Loss During Delivery
Acronym: QUOTABL
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Rachana Gavara, Assistant Professor of Obstetrics and Gynecology, Columbia University
Other Study IDs: AAAR4466
Record Dates: First submitted 2017-07-26; First posted 2017-07-28 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Hemorrhage, Postpartum
Keywords: Postpartum; Hemoglobin
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Antepartum Patients: Includes antepartum patients receiving prenatal care at the Broadway Practice who plan to deliver at Allen Hospital in New York City (NYC). On postpartum day 1 and day 2, a sample of blood will be drawn in the morning for hemoglobin and hematocrit estimation.
  Interventions: Procedure: Blood Draw

INTERVENTIONS:
Procedure: Blood Draw — On postpartum day 1 and day 2, a sample of blood will be drawn in the morning for hemoglobin and hematocrit estimation.

SUMMARY:
This is a prospective cohort study of patients delivering at Columbia University Medical Center/ Allen Hospital. For the primary research question, the investigators will compare the change in maternal hemoglobin from postpartum day 1 to day 2 and also determine correlation with estimation of blood loss (EBL) and quantitative blood loss (QBL).

DETAILED DESCRIPTION:
Postpartum hemorrhage is a leading cause of maternal mortality and morbidity worldwide. Early intervention is dependent on care providers ability to accurately estimate ongoing blood loss. Studies in the past have shown that obstetricians and midwives tend to overestimate blood loss when the lost volumes are small while tend to underestimate by as much as 40 to 50 percent when a large volume of blood is lost.

Multiple studies have shown that routine hemoglobin assessment in postpartum patients after uneventful delivery either vaginal or via cesarean section, is not necessary. This leads to increased cost of care without any added benefit and causes inconvenience to the patients. However knowing how imprecise blood loss estimation can be it is reasonable to screen women for anemia prior to discharge.

ELIGIBILITY:
Inclusion Criteria:

All antepartum patients receiving prenatal care at the Broadway Practice and plan to deliver at Allen Hospital in NYC.

Exclusion Criteria:

Patients who gave consent to participate in the study but did not deliver at Allen hospital.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women who are admitted to the Allen hospital for delivery during the recruitment period.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2019-01-04 (Actual); Study Completion 2019-04-23 (Actual)

PRIMARY OUTCOMES:
Change in maternal hemoglobin | Day 1 and Day 2
  Maternal hemoglobin will be measured on postpartum day 1 to day 2
Correlation of maternal hemoglobin to EBL | Up to 2 days after delivery
  Maternal hemoglobin will be measured to assess correlation to visually estimated blood loss
Correlation of maternal hemoglobin to QBL | Up to 2 days after delivery
  Maternal hemoglobin will be measured to assess correlation to quantified blood loss

CONTACTS AND LOCATIONS:
Overall Officials: Rachana Gavara, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No plans for sharing as this is a pilot study.